CLINICAL TRIAL: NCT02875613
Title: An Open-label, Single-arm, Multi-institutional Phase II Trial of Avelumab for Recurrent, Metastatic Nasopharyngeal Carcinoma
Brief Title: Avelumab for Recurrent/Metastatic Nasopharyngeal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow patient accrual
Sponsor: Assuntina Sacco, M.D. (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Assuntina Sacco, M.D., Assistant Professor, Medicine, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 160114
Record Dates: First submitted 2016-08-18; First posted 2016-08-23 (Estimated); Results first posted 2019-09-06 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Nasopharyngeal Cancer
Keywords: Nasopharyngeal; PD-L1; monoclonal antibody; Epstein-barr virus
MeSH Terms: conditions — Nasopharyngeal Neoplasms; Epstein-Barr Virus Infections | interventions — avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Avelumab (Experimental): Avelumab 10mg/kg IV infusion on days 1 and 15 of 28-day cycle
  Interventions: Drug: Avelumab

INTERVENTIONS:
Drug: Avelumab — Avelumab 10mg/kg IV on days 1 and 15 of each 28-day cycle. Treatment will be given until disease progression, unacceptable toxicity, investigator decision or patient withdrawal.
  Other Names: MSB0010718C

SUMMARY:
The purpose of this study is to determine whether avelumab, an investigational antibody against programmed death-ligand (PD-L1), has an effect on recurrent nasopharyngeal cancer. Avelumab is designed to block the interaction between programmed cell death protein 1 (PD-1), a known immune checkpoint, and PD-L1. By blocking this interaction, the immune system may be stimulated, allowing it to more effectively recognize and attack the cancer.

DETAILED DESCRIPTION:
This is a prospective, multi-center, open-label, single-arm phase II trial to evaluate the efficacy of Avelumab for patients with recurrent/metastatic, Epstein-Barr virus (EBV)-related nasopharyngeal carcinoma.

Upon study entry, all patients will receive Avelumab 10 milligrams per kilogram (mg/kg) intravenously (IV) on days 1 and 15 of each 28-day cycle. Treatment will be given until disease progression, unacceptable toxicity, investigator decision or patient withdrawal. Dose interruptions may occur per pre-specified criteria for grade 3 or higher toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patient has histologically/cytologically confirmed, non-keratinizing/undifferentiated, EBV-related nasopharyngeal carcinoma, not amenable to curative intent therapy. EBV testing may be completed per institutional standards.
* Patient must have at least one measurable site of disease as defined by RECIST v1.1, determined by investigator review
* Patient has received at least one prior line of systemic therapy in the recurrent/metastatic setting
* Patient is willing to undergo a fresh tumor biopsy (core or excisional) for correlative analyses (ie. PD-L1 expression).The study chair may grant exceptions to the mandatory biopsy should the treating physician deem that a biopsy is not feasible or unsafe for the patient, and archival tissue is available and provided for study purposes. A conversation with the study chair is required to obtain an exception.
* Patient has adequate organ and marrow function.
* Female patient of childbearing potential has a negative serum or urine pregnancy within 72 hours prior to receiving the first dose of study medication

Exclusion Criteria:

* Patient is currently receiving or has received another investigational agent within 4 weeks prior to Day 1 of study.
* Patient has received chemotherapy or radiotherapy within 4 weeks prior to Day 1 of study. Prior palliative radiotherapy to metastatic lesion(s) is permitted, provided there is at least one measurable lesion that has not been radiated.
* Patient has received prior immunotherapy with inhibitors of PD-1/PD-L1 axis.
* Patient has had major surgery or insufficient recovery from surgical-related trauma or wound healing within 14 days of Study Day 1.
* Patient has had a prior Grade ≥ 3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE > Grade 1.
* Patient has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Patient has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Patient has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs).Patients with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment within the past 2 years are not excluded.Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Patient has a diagnosis of immunodeficiency, or is receiving systemic steroid therapy (>10mg prednisone daily, or steroid equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of avelumab.
* Patient has a known history of active TB (Bacillus Tuberculosis).
* Patient has a known history of, or any evidence of active, non-infectious pneumonitis.
* Patient has a known history of chronic interstitial lung disease.
* Patient has an active infection requiring systemic therapy.
* Patient is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial.
* Patient has known active Hepatitis B infection (defined as presence of HepB sAg and/ or Hep B DNA), active hepatitis C infection (defined as presence of Hep C RNA) and/or known Human Immunodeficiency Virus (HIV). Patients with HIV who have a normal CD4 count (≥ 200) and an undetectable viral load are not excluded.
* Patient has received a live vaccine within 30 days of study Day 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2019-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Assuntina Sacco, MD, Principal Investigator — University of California Medical Center
Locations (2):
- United States (2):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Description of discrepancy between the enrollment number in the Protocol Section (6) and number of participants Started in the Participant Flow module (5): there were a total of six participants who signed consent for the study. One of the participants was a screen fail. Another participant withdrew consent prior to completing screening procedures. When determining the number of participants enrolled, these two participants were still considered. The correct enrollment number should be four.
Period: Overall Study
Arm/Group | Avelumab
Started | 6
Completed | 4
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Screen Failure | 1

BASELINE CHARACTERISTICS:
Arm/Group | Avelumab
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.25 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Based on Response Evaluation Criteria in Solid Tumors (RECIST)
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab
Number analyzed (Participants) | 4
Participants
  Progressive Disease at 6 months | 2
  Stable Disease at 6 months | 2

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Avelumab
All-Cause Mortality (participants affected / at risk) | 2/4
Serious Adverse Events (participants affected / at risk) | 3/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Avelumab (N=4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Blood bilirubin increased (Investigations) | 1
Hepatic hemorrhage (Hepatobiliary disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Sepsis (Infections and infestations) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Avelumab (N=4)
Hyponatremia (Metabolism and nutrition disorders) | 2
Fever (General disorders) | 1
Chills (General disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Peritoneal infection (Infections and infestations) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Hepatic hemorrhage (Hepatobiliary disorders) | 1
Pain (General disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Skin infection (Infections and infestations) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Edema limbs (General disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Weight loss (Investigations) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Body odor (Skin and subcutaneous tissue disorders) | 1
Papulopustular rash (Infections and infestations) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Tooth infection (Infections and infestations) | 1
Pruritis (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-17): https://cdn.clinicaltrials.gov/large-docs/13/NCT02875613/Prot_SAP_000.pdf